CLINICAL TRIAL: NCT02852538
Title: An Innovative Family Based Treatment for Adults With Anorexia Nervosa Using Insights From Neurobiology
Brief Title: Outcomes of a Skill-Based Program for Eating Disorders
Acronym: NEW FED TR
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Eating Disorders Association (Other)
Responsible Party: Principal Investigator, Christina Wierenga, Associate Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110659
Record Dates: First submitted 2016-07-26; First posted 2016-08-02 (Estimated); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NEW FED TR for Anorexia (Experimental): NEW FED TR
  Interventions: Behavioral: NEW FED TR

INTERVENTIONS:
Behavioral: NEW FED TR — NEW FED TR is a five day treatment for adults with anorexia nervosa. It is a neurobiologically informed, interactive, family-based treatment that draws upon the specific etiological traits characterizing anorexia nervosa. It stands for Neurobiological research findings Enhanced With Family/Friends of those with Eating Disorders, addressing Trait Responses that both create a vulnerability to the illness and serve as markers for recovery through treatment (formerly reported as Temperament-Based Treatment).
  Other Names: Intensive Temperament Based Treatment

SUMMARY:
This study aims to measure the effect of a neurobiologically-guided intensive family based treatment for adults with anorexia nervosa.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of anorexia nervosa
* Illness onset at least 2 years prior to study
* Medically stable
* Identified carer to participate in treatment with participant

Exclusion Criteria:

* Developmental or intellectual disorder
* Diagnosis of substance abuse or dependence in 3 months prior to study
* Current suicidal thoughts
* Severe comorbid psychiatric disorder (e.g., psychotic disorder, bipolar disorder)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-02; Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index | 3 months post-treatment

SECONDARY OUTCOMES:
Eating Disorder Examination Total Score | 3 months post-treatment
  Clinical symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Christina Wierenga, PhD, Principal Investigator — University of California, San Diego; Laura Hill, PhD, Study Chair — The Center for Balanced Living
Locations (2):
- United States (2):
  - University of California San Diego, San Diego, California
  - The Center for Balanced Living, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Knatz S, Wierenga CE, Murray SB, Hill L, Kaye WH. Neurobiologically informed treatment for adults with anorexia nervosa: a novel approach to a chronic disorder. Dialogues Clin Neurosci. 2015 Jun;17(2):229-36. doi: 10.31887/DCNS.2015.17.2/sknatz. PMID 26246796
- [Background] Kaye WH, Wierenga CE, Knatz S, Liang J, Boutelle K, Hill L, Eisler I. Temperament-based treatment for anorexia nervosa. Eur Eat Disord Rev. 2015 Jan;23(1):12-8. doi: 10.1002/erv.2330. Epub 2014 Nov 6. PMID 25377622
- [Derived] Hill L, Peck SK, Wierenga CE, Kaye WH. Applying neurobiology to the treatment of adults with anorexia nervosa. J Eat Disord. 2016 Dec 5;4:31. doi: 10.1186/s40337-016-0119-x. eCollection 2016. PMID 27980771
- See also: UCSD Eating Disorder Treatment and Research Program — http://eatingdisorders.ucsd.edu